CLINICAL TRIAL: NCT05648019
Title: CD19-Directed Chimeric Antigen Receptor (CAR) T-Cell Therapy for Relapsed/Refractory B-Lineage Leukaemia / Lymphoma - A Feasibility Protocol
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHCELL18P1
Record Dates: First submitted 2022-08-01; First posted 2022-12-13 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Lymphoblastic Leukemia; Lymphoblastic Leukemia in Children; Lymphoblastic Leukemia, Acute Adult; B-cell Acute Lymphoblastic Leukemia; Large B-cell Lymphoma; CAR
Keywords: CAR T-cell therapy; Relapse/Refractory; B-ALL; B-Lineage Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CD19-directed CAR T-cell therapy for relapsed/refractory B-lineage leukaemia/lymphoma.
  Interventions: Biological: Anti-CD19 CAR T-cells

INTERVENTIONS:
Biological: Anti-CD19 CAR T-cells — A target per-protocol dose of vi able CD19 CAR transduced T-cells will consist of a single infusion of 0.2 to 5.0 x 10e6 lentiviral-transduced viable 41BB-CD19 CAR T-cells per kg body weight.

SUMMARY:
The purpose of this study is to describe feasibility of delivering point-of-care manufactured CD19-directed CAR T-cell therapy to patients with relapsed/ refractory B-lineage leukaemia/ lymphoma.

DETAILED DESCRIPTION:
This is a single arm, open-label, multi-center, phase II feasibility study to deliver point-of-care manufactured CD19-directed CAR T-cell therapy to patients with relapsed / refractory B-lineage leukaemia / lymphoma.

The study consists of the following phases:

1. Screening phase: Eligibility; enrolment
2. Preparatory phase: Bridging therapy (if required); leukapheresis; CAR T manufacturing; lymphodepletion.
3. Treatment phase: Infusion of single dose of anti-CD19 CAR T-cells
4. Follow-up Phase: Efficacy and safety monitoring up to 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Eligible disease conditions:

   1. Relapsed or refractory B-cell ALL (all must be satisfied)

      * Presence of lymphoblasts in bone marrow aspirate by morphologic assessment or positive minimal residual disease at screening.
      * Relapsed or refractory or ineligible for HSCT
      * For relapsed B-ALL: Documentation of CD19 tumour expression (e.g. by flow cytometry) demonstrated in bone marrow or peripheral blood within 3 months of study entry
   2. Relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma.
2. Age at screening:

   1. < 18 years (paediatric group); or
   2. ≥ 18 years (adult group)
3. Adequate organ functions:
4. Life expectancy more than 12 weeks.
5. Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening.
6. Must meet the institutional criteria to undergo leukapheresis or have a leukapheresis product of non-mobilized cells received and accepted by the manufacturing site.

Exclusion Criteria:

Patients with any of the following will be excluded:

* B-ALL with isolated extramedullary disease relapse
* Patients with concomitant genetic syndrome: such as patients with Fanconi anaemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down syndrome will not be excluded.
* Patients with Burkitt's lymphoma/leukaemia (i.e. patients with mature B-cell ALL; leukaemia with B-cell [sIg positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
* Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening
* Human Immunodeficiency Virus (HIV) positive test within 8 weeks of screening
* Presence of grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD)
* Active CNS involvement by malignancy, defined by CNS-3 per NCCN guidelines. Subjects with CNS-2 involvement or with history of CNS disease that have been actively treated are eligible.
* Patient has an investigational medicinal product within the last 30 days prior to screening.
* Pregnant or nursing women.
* Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants, unless they are using highly effective methods of contraception for a period of 1 year after the CAR T-cell infusion. All female patients of childbearing potential must have a negative pregnancy test performed within 48 hours before infusion of CAR T-cells.

The following are not strictly exclusion criteria but must be discussed with PI/Site-PI:

* Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
* Treatment with any prior gene therapy product
* Has had treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Protocol Feasibility | 3 years
  To describe feasibility of delivering point-of-care manufactured CD19-directed CAR T-cell therapy to patients with relapsed / refractory B-lineage leukaemia / lymphoma by assessing number and percentage of enrolled patients who have successful manufacturing of CAR T-cell product, and number and percentage of enrolled patients who go on to receive the CAR T-cell product.

SECONDARY OUTCOMES:
Overall Response Rate | 6 months
  To evaluate percentage of patients with complete response or partial response at 28 days, 3 months and 6 months post-infusion of the CD19-directed CAR T-cells.
Toxicity Evaluations | 6 months
  To evaluate overall incidence (percentage of infused patients) of toxicities post-infusion of CAR T-cells, in particular cytokine release syndrome (CRS) and neurotoxicity, and percentage with Grade 3 and above CRS and neurotoxicity following ASTCT definition and severity grading, and other toxicities as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shui Yen Soh, MD, Principal Investigator — KK Women's and Children's Hospital; Aloysius Ho, MD, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided